CLINICAL TRIAL: NCT03494634
Title: Study of Chidamide as a Single-agent Treatment for Patients With Recurrent and Metastatic Epstein-Barr Virus (EBV)-Associated Solid Tumors
Brief Title: Chidamide for Patients With Recurrent and Metastatic Epstein-Barr Virus (EBV)-Associated Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, director, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-Q08
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Experimental Tumor
MeSH Terms: conditions — Neoplasms, Experimental | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide (Experimental)
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide — Chidamide 30mg orally BIW. Treatment cycles are repeated every 4 weeks.

SUMMARY:
Study of Chidamide as a Single-agent Treatment for Patients With Recurrent and Metastatic Epstein-Barr virus (EBV)-associated Solid Tumors

DETAILED DESCRIPTION:
Chidamide，a novel histone deacetylase inhibitor has been approved for the treatment of relapsed or refractory peripheral T-cell lymphoma in China. The aim of this study was to observe the efficacy and safety of Chidamide as a single-agent treatment in patients with recurrent and metastatic Epstein-Barr virus (EBV)-associated solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as recurrent and metastatic Epstein-Barr virus (EBV)-associated solid tumors, including nasopharyngeal carcinoma and other solid tumors (Lymphoma excluded). Patients must have failed at least one systemic treatment and been refractory to platinum-containing regimens;
2. At least one measurable lesion according to criteria RECIST v1.1;
3. Age 18-70 years, male or female;
4. ECOG performance status 0-2;
5. Life expectancy no less than 3 months;
6. Adequate hepatic, renal and bone marrow function;
7. History of brain metastasis is eligible, but maintenance of hormone is not required;
8. Contraception during and 4 weeks after the study for patients at child bearing age;
9. Patients have signed the Informed Consent Form.

Exclusion Criteria:

1. Women during pregnancy or lactation, or fertile women unwilling to take contraceptive measures;
2. QTc elongation with clinical significance ( male˃ 450ms, female˃ 470ms), ventricular tachycardia, atrial fibrillation, cardiac conducting blockage, myocardial infarction within 1 year, congestive heart failure, symptomatic coronary heart disease that requires treatment;
3. pericardial effusion ≥10mm sum of echo-free spaces by echocardiography;
4. Patients have undergone organ transplantation;
5. Patients received symptomatic treatment for bone marrow toxicity within 7 days prior to enrollment;
6. Patients with active hemorrhage;
7. Patients with or with history of thrombosis, embolism, cerebral hemorrhage, or cerebral infarction;
8. Patients with active HBV or HCV infection;
9. continuous fever within 14 days prior to enrollment;
10. Had major organ surgery within 6 weeks prior to enrollment;
11. Impaired liver function ( Total bilirubin ˃ 1.5 times of normal maximum, ALT/AST˃ 2.5 times of normal maximum, for patients with infiltrative liver disease ALT/AST ˃ 5 times of normal maximum), impaired renal function (serum creatinin˃ 1.5 times of normal maximum);
12. Patients with mental disorders or those do not have the ability to consent;
13. Patients with drug abuse, long term alcoholism that may impact the results of the trial;
14. Patients who received treatment of HDAC inhibitors;
15. Non-appropriate patients for the trial according to the judgment of the investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2018-04-15 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate（ORR） | up to 2 years
  the total proportion of patients with complete response（CR）and partial response（PR）

SECONDARY OUTCOMES:
Disease Control Rate （DCR） | up to 2 years
  the total proportion of patients with complete response（CR）, partial response（PR）and Stable Disease（SD）
Duration of Response （DOR） | up to 2 years
  Time from first documented complete response (CR) or partial response (PR) until time of progression.
progression-free survival（PFS） | 2 years
  Time from treatment until disease progression or death
overall survival（OS） | 2 years
  Time from treatment until death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center of Sun Yat-Sen University (CCSU), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No